CLINICAL TRIAL: NCT03798015
Title: Neurologic Outcome After Mitral Valve Surgery
Status: Withdrawn | Type: Observational
Why Stopped: resource issues on site
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-02143; ch18Grapow3
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Mitral Valve Reconstruction
Keywords: mitral valve surgery; mitral valve stenosis; mitral valve insufficiency; minimal invasive mitral valve surgery; neurological outcome
MeSH Terms: conditions — Mitral Valve Stenosis; Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mitral valve surgery: outcome of mitral valve surgery (stroke yes or no)
  Interventions: Other: mitral valve surgery

INTERVENTIONS:
Other: mitral valve surgery — assessment of ischemic or hemorrhagic stroke subsequent to mitral valve surgery

SUMMARY:
Reconstructive mitral valve surgery is increasingly done by minimal- invasive anterolateral thoracotomy technique in contrast to surgical approach by sternotomy. The minimal invasive approach is favourable regarding surgical trauma, length of hospital stay and amount of blood loss.

This study is to investigate the neurological outcome after minimal- invasive mitral valve surgery compared to open mitral valve surgery by sternotomy.

Pre-, intra- and postsurgical data from mitral valve surgery derived from the Basel mitral valve registry (collected from 2009 until now) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* surgery for mitral valve (reconstruction or replacement) (maybe combined with surgery for tricuspid valve and/ or surgery for atrial septal defects and/or patent foramen ovale)

Exclusion Criteria:

* other surgical interventions then the surgical interventions mentioned in the inclusion criteria
* pre- existing neurological deficit; neurologic limitation in daily life
* emergency surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing a surgical mitral valve reconstruction or replacement at the University Hospital Basel from 2009 until today
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
occurence of stroke (yes/ no) subsequent to mitral valve surgery | post surgical from day of surgery until day of discharge from hospital (approx. 2 weeks)
  assessment of ischemic or hemorrhagic stroke subsequent to mitral valve surgery

CONTACTS AND LOCATIONS:
Overall Officials: Martin Grapow, Prof. Dr. MD, Principal Investigator — Klinik für Herzchirurgie, Universitätsspital Basel
Locations (1):
- Herzchirurgie University Hospital Basel, Basel, Switzerland